CLINICAL TRIAL: NCT02274688
Title: A Comparative Effectiveness Trial of Optimal Patient-Centered Care for US Trauma Care Systems
Brief Title: A Comparative Effectiveness Trial of Optimal Patient-Centered Care
Acronym: TSOS 5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 46615-EJ; IH-1304-6319 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2013-12-17; First posted 2014-10-24 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Post Traumatic Concerns; Post Traumatic Stress Disorder; Depression and Suicide Ideation; Alcohol and Drug Use
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Patient-centered care transition intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care - Nurse Notification of Patient Concerns (No Intervention): Randomized and will be blindly assessed.
- Patient-centered care transition (Experimental): Case management, information technology/mHealth innovations, stepped-up psychopharmacology and psychotherapy elements.
  Randomized and will be blindly assessed.
  Interventions: Behavioral: Stepped Care Management

INTERVENTIONS:
Behavioral: Stepped Care Management — Case management, information technology/mHealth innovations, stepped-up psychopharmacology and psychotherapy elements.
  Other Names: Intervention
  Arms: Patient-centered care transition

SUMMARY:
The nation's trauma care system, which includes trauma center hospitals & emergency departments, is where over 30 million Americans receive care after traumatic injuries each year. Injury victims are diverse patients who suffer from complications of the initial injury as well as from multiple complex medical & mental health conditions. Currently, high-quality patient-centered care is not the standard of care throughout US trauma care systems. Injured trauma survivors treated in trauma care systems frequently receive fragmented care that is not coordinated across hospital, emergency department, outpatient, & community settings. Post-injury care is frequently not individualized to integrate the patient's most pressing post-traumatic concerns & preferences into medical decision making. The investigators, as a group of front-line trauma center providers, patients, researchers & policy makers, have been working together for over a decade to integrate patient-centered care into US trauma care systems. The investigators began this work by asking groups of injured patients the key patient-centered question: "Of everything that has happened to you since your injury, what concerns you the most?" The investigators developed scientifically sound assessment tools that allowed us to follow patient concerns after injury hospitalization. In May of 2011, the investigators convened an American College of Surgeons' policy summit that addressed mental health & patient-centered care integration across US trauma care systems. As part of this policy summit, patient members of our team presented their experiences of traumatic injury & recovery. While giving injured patients a "voice" at the summit, these narratives did not move surgical policy makers to develop mandates or guidelines for patient-centered care. In contrast, presentations that included information from randomized comparative effectiveness trials & standardized outcome assessments convinced surgical policy makers to develop US trauma care system policy mandates & best practice guidelines for post-traumatic stress disorder & alcohol use problems. Our team now realizes that in order to optimally integrate patient-centered care into US trauma care systems, the investigators must use the best scientific methods that capture the highest-quality data. This PCORI proposal aims to demonstrate that a patient-centered care management treatment that addresses patient's post-injury concerns & integrates patient concerns & preferences into medical decision making, while also coordinating care, can improve outcomes of great importance to patients & their caregivers, front-line providers & policy makers. This proposal directly addresses two PCORI patient-centered research questions: "After a traumatic injury, what can I do to improve the outcomes that are most important to me?" & "How can front-line providers working in trauma care systems help me make the best decisions about my post-injury health & health care?"

ELIGIBILITY:
Inclusion Criteria:

* Seen in acute care emergency department or trauma center setting for injury
* At least three post traumatic concerns
* AND One of the following PTSD Checklist Score (PCL-C) greater than or equal to 35 Patient Health Questionnaire 9 - greater than or equal to 10 Any endorsement of suicidal ideation on the PhQ-9 Item 9

Exclusion Criteria:

* Non-English speaking
* Under 14 years of age
* Incarcerated
* Psychotic behavior
* Suffered head, spinal cord, or other severe injuries that prevent participation in the inpatient ward interview.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Prater L, Bulger E, Maier RV, Goldstein E, Thomas P, Russo J, Wang J, Engstrom A, Abu K, Whiteside L, Knutzen T, Iles-Shih M, Heagerty P, Zatzick D. Emergency Department and Inpatient Utilization Reductions and Cost Savings Associated With Trauma Center Mental Health Intervention: Results From a 5-year Longitudinal Randomized Clinical Trial Analysis. Ann Surg. 2024 Jan 1;279(1):17-23. doi: 10.1097/SLA.0000000000006102. Epub 2023 Sep 25. PMID 37747970
- [Derived] Whiteside LK, Vrablik MC, Russo J, Bulger EM, Nehra D, Moloney K, Zatzick DF. Leveraging a health information exchange to examine the accuracy of self-report emergency department utilization data among hospitalized injury survivors. Trauma Surg Acute Care Open. 2021 Jan 28;6(1):e000550. doi: 10.1136/tsaco-2020-000550. eCollection 2021. PMID 33553651
- [Derived] Zatzick D, Russo J, Thomas P, Darnell D, Teter H, Ingraham L, Whiteside LK, Wang J, Guiney R, Parker L, Sandgren K, Hedrick MK, Van Eaton EG, Jurkovich G. Patient-Centered Care Transitions After Injury Hospitalization: A Comparative Effectiveness Trial. Psychiatry. 2018 Summer;81(2):141-157. doi: 10.1080/00332747.2017.1354621. Epub 2018 Mar 13. PMID 29533154

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Usual Care - Nurse Notification of Patient Concerns: Randomized, nurse notified of high levels of psychological distress.
  Will be blindly assessed.
- Patient-centered Care Transition: Randomized, case management, information technology/mHealth innovations, stepped-up psychopharmacology and psychotherapy elements.
  Will be blindly assessed.
Period: Overall Study
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Started | 86 | 85
Completed | 72 | 72
Not Completed | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 74 | 77 | 151
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (16) | 41.2 (16.1) | 42.4 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 50 | 97
  Male | 39 | 35 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 80 | 76 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 5 | 15
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 5
  Black or African American | 13 | 8 | 21
  White | 51 | 47 | 98
  More than one race | 5 | 10 | 15
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 86 | 85 | 171

OUTCOME MEASURES:

1. Primary Outcome: Change in Post Traumatic Concerns Over the Course of the Six Months After Injury
Description: The primary outcome is the endorsement of ≥1 severe posttraumatic concerns.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
Participants
  Baseline | 80 | 83
  1-month | 55 | 59
  3-month | 45 | 48
  6-month | 42 | 33
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; Mixed Model Regression; Data from all 171 patients at all time points used in this intent-to-treat analytic approach. We hypothesize intervention patients will demonstrate diminished outcome severity over time when compared to nurse notification patients, as evidenced by a significant group by time interaction effect; Test type: Superiority; p = 0.01, Wald Chi-Square=11.29, df=3, P=0.01

2. Primary Outcome: Change in Post Traumatic Stress Disorder (PTSD) Symptoms Over the Course of the Six Months After Injury
Description: The investigators used the PTSD Checklist - Civilian (PCL-C) as a continuous measure. The scoring of the scale ranges from a minumum of 17 to a maximum of 85, with higher scores indicating a worse outcome. No subscales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
units on a scale
  Baseline | 42.9 (11.2) | 42.5 (11.3)
  1-month | 41.7 (14.3) | 43.7 (14.9)
  3-month | 40.7 (14.7) | 38.7 (13.7)
  6-month | 39.3 (14.7) | 38.6 (16.0)
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.23, Wald Chi-Square=3.01, df=3, p=0.23

3. Primary Outcome: Change in Depression Symptoms Over the Course of the Six Months After Injury
Description: The investigators used the Patient Health Questionnaire (PHQ-9) as a continuous measure, with scores ranging from 1 to 27. Higher scores represent a worse outcome. No subscales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patient-centered Care Transition: Case management, information technology/mHealth innovations, stepped-up psychopharmacology and psychotherapy elements.
  Stepped Care Management: Case management, information technology/mHealth innovations, stepped-up psychopharmacology and psychotherapy elements.
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
units on a scale
  Baseline | 14.8 (4.2) | 14.3 (4.5)
  1-month | 12.1 (6.2) | 13.2 (6.5)
  3-month | 11.7 (7.2) | 10.8 (6.9)
  6-month | 10.7 (6.4) | 9.3 (6.8)
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.23, Wald Chi-Square=4.25, df=3, p=0.23

4. Secondary Outcome: Alcohol Use Problems
Description: The investigators used the Alcohol Use Disorders Identification Test (AUDIT) as a continuous measure. The 10-item scale score ranges from 0-40, with higher values indicating a worse outcome. No sub scales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
units on a scale
  Baseline | 3.7 (3.2) | 3.4 (3.2)
  1-month | 1.1 (2.6) | 0.5 (1.6)
  3-month | 1.7 (2.8) | 1.1 (1.9)
  6-month | 2.3 (2.9) | 1.6 (2.5)
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.55, Wald Chi-Square=2.12, df=3, p=0.55

5. Secondary Outcome: Functional Status
Description: The investigators used the Medical Outcomes Study Short Form healthy survey (MOS SF-12/36) physical components summary to assess physical function. The minimum and maximum scores are 0-100 with higher scores representing a better outcome. No other subscales will be used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
units on a scale
  Baseline | 48.4 (9.1) | 48.5 (9.2)
  1-month | 38.3 (10.4) | 37.1 (10.9)
  3-month | 39.3 (9.9) | 39.8 (8.0)
  6-month | 39.9 (9.9) | 42.3 (8.4)
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.32, Wald Chi-Square=3.52, df=3; p=0.32

6. Secondary Outcome: Number of Participants With Suicidal Ideation
Description: The investigators used PHQ-9 item 9 to assess suicidal ideation. For the analysis, a score of > 0 on item 9 of PHQ-9 was considered a positive endorsement and a worse outcome.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
Participants
  Baseline | 19 | 22
  1-month | 13 | 18
  3-month | 21 | 14
  6-month | 16 | 17
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.26, Wald Chi-Square=4.02, df=3, p=0.26

7. Secondary Outcome: Number of Patients Carrying a Weapon
Description: The investigation used a single yes/no item to assess whether the patient was carrying a weapon.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
Participants
  Baseline | 7 | 12
  1-month | 4 | 3
  3-month | 7 | 5
  6-month | 5 | 9
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.22, Wald Chi-Square=4.44, df=3, p=0.22

8. Secondary Outcome: Number of Participants With One or More Emergency Department Visits Over Time
Description: The investigators used population level data on emergency department health service use for the intent-to-treat sample
Time Frame: The investigators assessed emergency department service use over the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
Participants
  Baseline | 41 | 44
  3-6 month | 26 | 14
  6-9 month | 27 | 18
  9-12 month | 26 | 19
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.08, Regression Poisson — F(3,507)=2.24, P=0.08

9. Secondary Outcome: Drug Use Problems
Description: The investigators used the Drug Abuse Screening Test (DAST-10) as a continuous outcome measure. DAST-10 scale scores range from 0 to 10, with higher scores representing a worse outcome. No subscales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
Number analyzed (Participants) | 86 | 85
units on a scale
  Baseline | 2.0 (1.9) | 2.2 (2.0)
  1-month | 1.4 (1.2) | 1.3 (1.2)
  3-month | 1.4 (1.4) | 1.3 (1.1)
  6-month | 1.3 (1.0) | 1.5 (1.4)
Statistical Analysis 1: Comparison: Enhanced Usual Care - Nurse Notification of Patient Concerns vs Patient-centered Care Transition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.36, Wald Chi-Square=3.24, df=3, p=0.36

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: Serious adverse event = Any documented suicide attempt Adverse event = Any PHQ-9, item 9, score >0
Arm/Group | Enhanced Usual Care - Nurse Notification of Patient Concerns | Patient-centered Care Transition
All-Cause Mortality (participants affected / at risk) | 0/86 | 2/85
Serious Adverse Events (participants affected / at risk) | 1/86 | 2/85
Other Adverse Events (participants affected / at risk) | 39/86 | 39/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care - Nurse Notification of Patient Concerns (N=86) | Patient-centered Care Transition (N=85)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enhanced Usual Care - Nurse Notification of Patient Concerns (N=86) | Patient-centered Care Transition (N=85)
PHQ-9 Score of >0 (Psychiatric disorders) | 39 | 39

LIMITATIONS AND CAVEATS:
Because this was a multifaceted intervention, the investigation did not yield information regarding which components of the treatment were effective in targeting specific outcomes. The intervention extended up until the 6-month injury time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No